CLINICAL TRIAL: NCT04118114
Title: An Open Label Phase II Study of the Efficacy and Tolerability of PRL3-ZUMAB and Predictive Biomarkers in Advanced Solid Tumours
Brief Title: Phase II Study of PRL3-ZUMAB in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: INTRA-IMMUSG PRIVATE LIMITED (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCS-2018-Phase2-PRL3
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer; Hepatocellular Carcinoma; Advanced Solid Tumor
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRL3-ZUMAB Monotherapy (Experimental)
  Interventions: Drug: PRL3-zumab

INTERVENTIONS:
Drug: PRL3-zumab — IV administration every 2 weeks

SUMMARY:
This is a Phase II, open-label, single dose level study of PRL3-ZUMAB monotherapy in patients with advanced solid tumours that have failed standard therapy. Approximately 30 patients will be recruited with ~10 gastric cancers and ~10 hepatocellular carcinomas. Patients who have received at least 1 dose of PRL3-ZUMAB will be evaluable for toxicity and efficacy.

PRL3-ZUMAB will be given IV every 2 weeks for up to 12 infusions in the absence of unmanageable toxicities or disease progression. Patients who are benefitting from the treatment may continue on PRL3-ZUMAB beyond 12 infusions with the agreement of the study drug provider.

PRL3-ZUMAB at the RP2D in tumour types enriched for known PRL-3 expression for efficacy and tolerability will be evaluated. There will also be in depth molecular profiling of tissues in patients who have an objective response or prolonged disease stabilization to identify predictive/selection biomarkers as well as evaluation of the oncogenic signaling modulation and immunomodulation by PRL3-ZUMAB and its potential for future combination with other targeted therapies or immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 21 years of age or older at the time written informed consent is obtained.
* Histopathological- or cytological- documented advanced curatively unresectable solid tumors failing standard therapy.

  * For HCC must have failed at least 1 line of standard therapy.
  * For gastric cancer must have failed at least 2 line of standard therapy (inclusive of adjuvant treatment).
  * For other solid tumours must have failed at least 1 line of standard therapy.
* Progressive disease following the last treatment
* Life expectancy ≥ 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status (ECOG PS) score of ≤ 2 at study entry
* Recovery to Grade ≤ 1 by the Common Terminology Criteria for Adverse Events, Version 4.03 (CTCAE v 4.03), from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies for cancer, with the exception of non-clinically significant adverse events such as alopecia; biochemical abnormalities, or resolved to Grade ≤ 2: peripheral neuropathy; hypertension and proteinuria.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at study entry. Subjects not considered WOCBP are those without menses for 24 consecutive months, and those who have undergone hysterectomy and/or bilateral salpingo-oophorectomy. WOCBP must be willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of the study.
* Adequate organ and hematological function as evidenced by the following laboratory studies within 10 days of 1st treatment:

  * Absolute neutrophil count ≥ 1.0 x 10^9/L.
  * Platelet count ≥ 75 x 10^9/L. Hemoglobin ≥ 9 g/dL.
  * Prothrombin time and activated partial thromboplastin time ≤ 1.5 x upper limit of normal (ULN) per institutional laboratory normal range.
  * Total bilirubin ≤ 1.5x ULN.
  * Aspartate aminotransferase and alanine aminotransferase ≤ 3 x ULN (≤ 5x ULN in the presence of liver mets).
  * For patients with hepatocellular carcinoma (HCC) Child Pugh score of ≤ B7.
  * Creatinine < 1.5x ULN
* Evaluable or measurable disease by RECIST v1.1
* Patients with active Hepatitis B (defined as Hep B S Ag or DNA positive) need to be on anti-viral therapy while on PRL3-ZUMAB.

Exclusion Criteria:

* Untreated or symptomatic central nervous system metastases. Patients with treated brain metastases stable for 3 months are eligible to enroll.
* Major surgical procedures within 28 days prior to enrolment.
* Pregnant or breast-feeding females.
* Known HIV infection.
* Treatment with any of the following anti-cancer therapies prior to the first dose of study drugs within the stated time frames:

  * Prior chemotherapy ≤ 2 weeks of C1 Day 1 of PRL3-ZUMAB.
  * Biological therapy (e.g., antibodies) within a period of time that is ≤ 5 t1/2 or ≤ 3 weeks, whichever is shorter, prior to starting study drug.
  * Continuous or intermittent small molecule therapeutics within a period of time that is ≤ 5 t1/2 or ≤ 3 weeks (whichever is shorter) prior to starting study drug.
  * Any other investigational agents within a period of time that is ≤ 5 t1/2 or less than the cycle length used for that treatment or ≤ 4 weeks (whichever is shortest) prior to starting study drug.
  * Wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug.
* Patients requiring regular immunosuppressive medication for autoimmune disease or corticosteroid doses of >10mg prednisolone for greater than 2 days
* Unable to provide informed consent.
* History of another cancer within the last 2 years, with the exception of

  * Curatively resected non-melanomatous skin cancer,
  * Curatively treated cervical carcinoma in-situ,
  * Prostate cancer treated with leuteinizing hormone-releasing hormone (LH-RH) agonists/pure antagonists for at least 2 months
* Prior stem cell or bone marrow transplant
* Vaccinated within 2 weeks from prior to the first administration of PRL3-ZUMAB

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From start of treatment to first occurence of disease progression or death, up to 2 years
Number of patients that do not have disease progression at 16 weeks from start of treatment | 16 weeks after start of treatment
  Clinical benefit rate at 16 weeks
Treatment related adverse events rate | From start of treatment to 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ng, MD, Principal Investigator — National Cancer Centre of Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thura M, Al-Aidaroos AQO, Yong WP, Kono K, Gupta A, Lin YB, Mimura K, Thiery JP, Goh BC, Tan P, Soo R, Hong CW, Wang L, Lin SJ, Chen E, Rha SY, Chung HC, Li J, Nandi S, Yuen HF, Zhang SD, Guan YK, So J, Zeng Q. PRL3-zumab, a first-in-class humanized antibody for cancer therapy. JCI Insight. 2016 Jun 16;1(9):e87607. doi: 10.1172/jci.insight.87607. PMID 27699276
- [Background] Guo K, Li J, Tang JP, Tan CP, Hong CW, Al-Aidaroos AQ, Varghese L, Huang C, Zeng Q. Targeting intracellular oncoproteins with antibody therapy or vaccination. Sci Transl Med. 2011 Sep 7;3(99):99ra85. doi: 10.1126/scitranslmed.3002296. PMID 21900592